CLINICAL TRIAL: NCT00379535
Title: Phase III : Preventing Lack of Iodine During Pregnancy. Effect of Supplying Woman With Potassium Iodine to the Neuro-Cognitive Children Development Until Two Years
Brief Title: Preventing Lack of Iodine During Pregnancy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0501101; PHRC
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Pregnancy
Keywords: pregnancy , lack of iodine; lack of iodine during pregnancy
MeSH Terms: interventions — Potassium Iodide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Daily dose of 200 µg of potassium iodide
  Interventions: Drug: potassium iodide
- 2 (Placebo Comparator): Daily dose of placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: potassium iodide — per os
  Other Names: Iodence
  Arms: 1
Drug: placebo — per os
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of potassium iodide during pregnancy on neuro-cognitive development of children followed up until two years.

DETAILED DESCRIPTION:
374 patients with pregnancy less 12 weeks amenorrhea

Patients randomized in 2 parallel groups (each group with 187 patients)

* one group with 200 µg of potassium iodide
* one group with placebo

Follow up during 3 years with :

* a selection visit, an inclusion with randomization before 12 weeks amenorrhea
* and follow up visit at the 5th month and 8th month of pregnancy, the day of birth, and 6, 12, and 24 months " post partum "

ELIGIBILITY:
Inclusion Criteria:

* Patients with pregnancy less 12 weeks amenorrhea , with clinically normal pregnancy, unique or twiny
* Patients who agree to take part in the study and able to sign an Informed Consent Form

Exclusion Criteria:

* Patients receiving a treatment for thyroid affection, or with thyroid pathology
* Patients with a chronic pathology like insulin dependent diabetes or arterial hypertension
* Patients with a treatment supplying iodine or having had a gynecologic exam with a iodine solution in the last 30 days
* Patients taking part in another clinical test or in the last 30 days
* Patients with depressive antecedent before pregnancy or taking antidepressant treatment
* Psychiatric troubles that may interfere with the clinical evaluation
* Patients under special supervision or trusteeship
* No social security cover

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 374 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Supplying a daily dose of 200 µg of potassium iodide in comparison with a placebo dose to pregnant woman and evaluate the impact on neuro-cognitive development of children followed up until two years | 2 years

SECONDARY OUTCOMES:
Prevalence of hypothyroxinemia and hypothyroidism during pregnancy | 9 months max
Change in the functional thyroid parameters of mother during iodine treatment | 2 years
Comparison of the psychometric development of children , for woman with and without treatment | 6, 12, and 24 months
Quantify the iodine supply from the woman to the baby during the breast feeding for woman with and without iodine treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: CARON PHILIPPE, Pr, Principal Investigator — University Hospital, Toulouse; WEMEAU Jean-Louis, Pr, Study Chair — CHRU LILLE; NICCOLI-SIRE Patricia, Pr, Study Chair — CHU Timone MARSEILLE; BRUCKER-DAVIS Francoise, Dr, Study Chair — CHU NICE
Locations (1):
- Endocrinology - University Hospital, Toulouse, France

REFERENCES:
- [Background] Caron P, Hoff M, Bazzi S, Dufor A, Faure G, Ghandour I, Lauzu P, Lucas Y, Maraval D, Mignot F, Ressigeac P, Vertongen F, Grange V. Urinary iodine excretion during normal pregnancy in healthy women living in the southwest of France: correlation with maternal thyroid parameters. Thyroid. 1997 Oct;7(5):749-54. doi: 10.1089/thy.1997.7.749. PMID 9349578
- [Background] Caron Ph, D Glinoer La fonction thyroïdienne au cours de la grossesse La Thyroïde. De la physiologie cellulaire aux dysfonctionnements. Des concepts à la pratique. Ed Expansion Scientifique - Paris, 2001, 495-500.